CLINICAL TRIAL: NCT02651155
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Lubiprostone for the Treatment of Chronic Idiopathic Constipation
Brief Title: Lubiprostone for the Treatment of Chronic Idiopathic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lubiprostone-3001; U1111-1170-0417 (Registry Identifier: WHO)
Record Dates: First submitted 2016-01-07; First posted 2016-01-08 (Estimated); Results first posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2017-11

CONDITIONS: Constipation
Keywords: Drug therapy
MeSH Terms: conditions — Constipation | interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lubiprostone 24 μg (Experimental): Lubiprostone 24 μg, capsules, orally, twice daily, under fed conditions, for 4 weeks.
  Interventions: Drug: Lubiprostone
- Placebo (Placebo Comparator): Lubiprostone placebo-matching capsules, orally, twice daily, under fed conditions, for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lubiprostone — Lubiprostone capsules
  Arms: Lubiprostone 24 μg
Drug: Placebo — Lubiprostone placebo-matching capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of oral administration of lubiprostone 24 μg twice daily (BID) for 4 weeks in participants with chronic idiopathic constipation (CIC) compared with placebo.

DETAILED DESCRIPTION:
The drug being tested in this study is called lubiprostone. Lubiprostone is being tested to treat people who have chronic idiopathic constipation. This study will look at the frequency of spontaneous bowel movements (SBMs) in people who take lubiprostone compared to placebo.

The study will enroll approximately 204 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups, such that equal numbers of subjects will be in each treatment group-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Lubiprostone 24 μg
* Placebo (dummy inactive pill) - this is a capsule that looks like the study drug but has no active ingredient

All participants will be asked to take one capsule with breakfast and one capsule with dinner each day throughout the study. All participants will be asked to record each time they have a SBM and all details of each SBM (including the consistency of the stool and the difficulty they have in passing it) in a diary.

This multi-center trial will be conducted in Russia. The overall time to participate in this study is 8 weeks. Participants will make multiple visits to the clinic, and will be contacted by telephone 14 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Has a history of constipation defined as having spontaneous bowel movement (SBM) frequency of less than 3 times per week on average for 6 months or longer and for whom the same SBM frequency is observed during the Screening Period.
4. Has had 1 or more of the symptoms associated with SBM (described below) for 6 months or longer at the start of Screening:

   1. Scybalum stool or hard feces in at least 1 out of every4 bowel movements.
   2. Sensation of incomplete evacuation in at least 1 out of every 4 bowel movements.
   3. Straining in at least 1 out of every 4 bowel movements.
5. Rarely has loose stools without the use of laxatives.
6. Is willing and able to keep a diary on his/her own and willing and able to complete a questionnaire.
7. Is male or female and aged 18 years or older, at the time of signing an informed consent.
8. A female participant of childbearing potential who is sexually active agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study and 14 days after the last dose of study drug.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to Screening.
2. Has received lubiprostone in a previous clinical study or as a therapeutic agent.
3. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. Has, in the judgment of the investigator, clinically significant abnormal hematological parameters of hemoglobin, hematocrit, or erythrocytes at Screening.
5. Has a history or clinical manifestations of significant mechanical obstruction (intestinal obstruction due to tumor, hernia etc).
6. Has a history of hypersensitivity or allergies to lubiprostone or any of its excipients.
7. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Screening Visit.
8. Is required to take excluded medications.
9. If female, is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
10. Participant whose constipation is considered to be due to drugs or to whom a prohibited concomitant medication has been administered.
11. Is having chronic constipation due to a secondary cause (medications, diabetes mellitus, hypothyroidism, depression, etc.)
12. Has sufficient criteria for irritable bowel syndrome (IBS) or functional defecation disorder.
13. SBM frequency is 3 or more per week.
14. SBM frequency has been less than 3 times per week for less than 6 months in duration or whose symptoms associated with SBM have been present for less than 6 months (hard feces, sensation of incomplete evacuation, or straining).
15. Received treatment with a rescue medication within 24 hours prior to the first dose on the morning of Day1: bisacodyl suppository, which is a standard laxative, glycerin enema, or any other rescue medication.
16. Has megacolon/megarectum or has received a diagnosis of intestinal pseudo-obstruction.
17. Has confirmed or suspected organic disorders of the large intestine (obstruction, stenosis, carcinoma, or inflammatory bowel disease). Organic disorders of the large intestine can be confirmed or ruled out using the results of enema X-ray examination or total colonoscopy performed in the previous 2 years. If the participant has no history or shows no current evidence of weight loss, anemia, or rectal bleeding, organic disorders may be ruled out based on the results of such testing performed in the past 3 years. Any participant in whom total colonoscopy has detected a polyp requiring treatment is excluded from this study .Note: Participant should not be screened unless at least 7 days have passed since an enema X-ray examination, total colonoscopy or sigmoidoscopy have been performed.
18. Has been hospitalized for gastrointestinal or abdominal surgery within 3 months prior to Screening.
19. Has a significant cardiovascular, liver, lung, kidney, neurological, or mental disease (including existing alcohol or drug abuse problem) or a systemic disease.
20. Has significant clinical findings or in whom a significant abnormality has been found in hematology test, serum chemistry, or urinalysis.
21. Participant in whom noncompliance with the study protocol (administration schedule, visit schedule, diary completion or other study procedure) is expected.
22. Has a history of malignant disease (except basal cell carcinoma) within 5 years prior to Screening.
23. Has any screening abnormal laboratory value that suggests a clinically significant underlying disease or condition that may prevent the participant from entering the study; or the participant has: creatinine >1.5 mg/dL, alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2 times the upper limit of normal (ULN), or total bilirubin >2.0 mg/dL with AST/ALT elevated above the limits of normal values.
24. Participant who the investigator/subinvestigator has determined ineligible to participate in this study for any reason other than the above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2017-01-11 (Actual); Study Completion 2017-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (12):
- Russia (12):
  - Saint Petersburg, Pushkin
  - Barnaul
  - Kazan'
  - Kemerovo
  - Krasnodar
  - Moscow
  - Novosibirsk
  - Omsk
  - Saint Petersburg
  - Samara
  - Ulyanovsk
  - Yaroslavl

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 20 investigative sites in Russia from 17 February 2016 to 26 January 2017.
Pre-assignment Details: Participants with a diagnosis of chronic idiopathic constipation as determined by the Rome III Diagnostic Criteria for Functional Constipation were enrolled in 1:1 ratio to receive lubiprostone or placebo.
Groups:
- Placebo: Lubiprostone placebo-matching capsules, orally, twice daily, for up to 4 weeks.
- Lubiprostone 24 μg: Lubiprostone 24 μg, capsules, orally, twice daily, for up to 4 weeks.
Period: Overall Study
Arm/Group | Placebo | Lubiprostone 24 μg
Started | 99 | 105
Completed | 93 | 103
Not Completed | 6 | 2
Not completed — Pretreatment Event/Adverse Event | 1 | 2
Not completed — Voluntary Withdrawal | 5 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized to receive study treatment whether or not they received treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lubiprostone 24 μg | Total
Number analyzed (Participants) | 99 | 105 | 204
Age, Continuous [Mean (Full Range); unit: years] | 49.0 [20 to 84] | 51.1 [19 to 79] | 50.1 [19 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 90 | 171
  Male | 18 | 15 | 33
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 1 | 1
  White | 99 | 102 | 201
  Multiracial | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Russia | 99 | 105 | 204
Height [Mean (Standard Deviation); unit: cm] | 166.2 (7.16) | 165.1 (7.77) | 165.6 (7.49)
Weight [Mean (Standard Deviation); unit: kg] | 70.08 (14.206) | 68.75 (11.240) | 69.39 (12.751)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.265 (4.2558) | 25.254 (4.0513) | 25.259 (4.1415)
Smoking Classification [Number; unit: participants]
  Participant has never smoked | 87 | 88 | 175
  Participant is a current smoker | 9 | 11 | 20
  Participant is an ex-smoker | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Spontaneous Bowel Movement (SBM) Frequency at Week 1
Description: A SBM is defined as any bowel movement (BM) that does not occur within 24 hours after rescue medication use (laxative, suppository, or enema). SBM frequency data was collected in a diary. Participants were given a diary to complete at home where they recorded the date and time of each BM.
Time Frame: Week 1
Population: FAS included all participants who were randomized to receive study treatment whether or not they received treatment. Missing values were imputed by last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: SBMs/week
Arm/Group | Placebo | Lubiprostone 24 μg
Number analyzed (Participants) | 99 | 105
SBMs/week | 3.6 (2.51) | 5.0 (2.94)
Statistical Analysis 1: Comparison: Placebo vs Lubiprostone 24 μg; Test type: Superiority or Other; p = 0.003, Van Elteren Test; SBM was analyzed using Van Elteren Test stratified by center. Centers with less participants were pooled based on geographical proximity; Median Values of CI = 1.0, 95% CI 2-sided [0.1 to 1.0] — CI was estimated by inverting the hypothesis test

2. Secondary Outcome: SBM Frequency at Weeks 2, 3 and 4
Description: A SBM is defined as any BM that does not occur within 24 hours after rescue medication use. SBM frequency data was collected in a diary. Participants were given a diary to complete at home where they recorded the date and time of each BM.
Time Frame: Weeks 2, 3 and 4
Population: FAS included all participants who were randomized to receive study treatment whether or not they received treatment. Missing values were imputed by LOCF method.
Measure: Mean (Standard Deviation); unit: SBMs/week
Arm/Group | Placebo | Lubiprostone 24 μg
Number analyzed (Participants) | 99 | 105
SBMs/week
  Week 2 | 3.9 (2.52) | 5.0 (2.82)
  Week 3 | 3.8 (2.87) | 5.1 (2.72)
  Week 4 | 3.7 (2.72) | 5.2 (2.61)

3. Secondary Outcome: Percentage of Participants Who Had a SBM Within 24 Hours After the First Dose of Study Medication
Description: A SBM is defined as any BM that does not occur within 24 hours after rescue medication use. Percentage of participants who had a SBM within 24 hours after the first dose was assessed and derived from the data on SBMs collected in the participant diary.
Time Frame: Up to 24 hours after the first dose of study medication
Population: FAS included all participants who were randomized to receive study treatment whether or not they received treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Lubiprostone 24 μg
Number analyzed (Participants) | 99 | 105
percentage of participants | 35.4 | 46.7

4. Secondary Outcome: Mean Degree of Straining Score
Description: For each participant, the mean degree of straining was averaged for all SBMs in a given week. The degree of straining for each SBM was collected in the participant diary. The degree of straining is scored on a 5-point scale where: 0=No straining, 1=Mild straining, 2=Moderate straining, 3=Strong straining or 4=Very strong straining with higher scores indicating more severe straining.
Time Frame: Weeks 1, 2, 3 and 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Lubiprostone 24 μg
Number analyzed (Participants) | 99 | 105
scores on a scale
  Week 1 | 2.3 (1.09) | 1.7 (1.01)
  Week 2 | 2.0 (1.11) | 1.6 (1.04)
  Week 3 | 1.9 (1.19) | 1.4 (0.99)
  Week 4 | 2.0 (1.19) | 1.3 (1.00)

5. Secondary Outcome: Mean Degree Stool Consistency Score
Description: For each participant, the mean stool consistency score was averaged for all SBMs in a given week. The mean degree of stool consistency for each SBM was collected in the participant diary based on the Bristol Stool Chart. The Bristol Stool Chart is a visual medical aid designed to classify the form of human feces into seven categories where: 1=Hard and round (difficult-to-pass), 2=Sausage-shaped but hard stool, 3=Sausage-shaped stool with cracks on the surface, 4=Sausage-shaped, soft stool with smooth surface, or coiled stool, 5=Soft, half-solid (and easy-to-pass) stool with clear crease, 6=Unshaped, loose stool with small, irregular-shaped pieces, or mushy stool or 7=Watery stool without solid pieces (entirely liquid).
Time Frame: Weeks 1, 2, 3 and 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Lubiprostone 24 μg
Number analyzed (Participants) | 99 | 105
scores on a scale
  Week 1 | 3.0 (1.10) | 3.6 (1.37)
  Week 2 | 3.3 (1.08) | 3.7 (1.33)
  Week 3 | 3.2 (1.11) | 3.8 (1.28)
  Week 4 | 3.0 (1.06) | 3.8 (1.30)

6. Secondary Outcome: Weekly Abdominal Symptoms Score
Description: The abdominal symptoms (bloating and discomfort upon waking in the morning) were scored weekly on a 5-point scale, where: 0=None, 1=Mild, 2=Moderate, 3=Severe or 4=Very severe, with a higher score indicating more severe symptoms. Assessment of weekly abdominal symptoms were recorded by the participant in the diary.
Time Frame: Weeks 1, 2, 3 and 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a sclae
Arm/Group | Placebo | Lubiprostone 24 μg
Number analyzed (Participants) | 99 | 105
scores on a sclae
  Abdominal Bloating, Week 1 | 1.6 (1.00) | 1.5 (0.86)
  Abdominal Bloating, Week 2 | 1.5 (1.04) | 1.3 (0.94)
  Abdominal Bloating, Week 3 | 1.6 (1.02) | 1.2 (1.01)
  Abdominal Bloating, Week 4 | 1.4 (1.03) | 1.1 (0.93)
  Abdominal Discomfort, Week 1 | 1.7 (0.98) | 1.5 (0.95)
  Abdominal Discomfort, Week 2 | 1.6 (1.07) | 1.3 (0.98)
  Abdominal Discomfort, Week 3 | 1.6 (1.06) | 1.2 (1.01)
  Abdominal Discomfort, Week 4 | 1.5 (1.02) | 1.2 (0.97)

ADVERSE EVENTS:
Time Frame: Baseline and up to Week 6
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Lubiprostone 24 μg
Serious Adverse Events (participants affected / at risk) | 1/99 | 0/105
Other Adverse Events (participants affected / at risk) | 6/99 | 16/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=99) | Lubiprostone 24 μg (N=105)
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=99) | Lubiprostone 24 μg (N=105)
Nausea (Gastrointestinal disorders) | 3 | 11
Diarrhoea (Gastrointestinal disorders) | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.